CLINICAL TRIAL: NCT02668081
Title: Prospective Randomized Study Comparing the Effects of Endoscopic Sphincterotomy (EST) and Endoscopic Papillary Balloon Dilation (EPBD) in Patients With Acute Biliary Pancreatitis (ABP)
Brief Title: Comparing the Effects of EST and EPBD in Patients With Acute Biliary Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Hoi-Hung Chan, associate professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS15-CT7-13
Record Dates: First submitted 2016-01-08; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Acute Biliary Pancreatitis
Keywords: Endoscopic sphincterotomy; Endoscopic papillary balloon dilation; Metagenomics
MeSH Terms: interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic papillary balloon dilation (Experimental): For EPBD group, after selective cannulation of the common bile duct by the catheter, cholangiography will be performed to confirm the diagnosis of bile duct pathology. A 0.025-0.035-inch guidewire will then be inserted into the bile duct through the catheter. A dilating balloon (The controlled radial expansion (CRE) balloon dilation catheter, CRE balloon 5.5 cm (centimeter) in length, 1-1.2 cm/1.2-1.5 cm/1.5-2.0 cm in diameter) will be passed via the pre-positioned guidewire into the bile duct. Using fluoroscopic and endoscopic guidance, the balloon will be inflated with contrast medium up to the optimal size and duration (normally 5min (minutes)) after the waist on the balloon disappeared according to the patients' condition and tolerance.
  Interventions: Procedure: Endoscopic papillary balloon dilation
- Endoscopic sphincterotomy (Active Comparator): For EST group,endoscopic sphincterotomy(EST) will be done as large as possible with a pull type sphincterotome (The TRUEtome, Biliary sphincterotomy sphincterotome, Single-use sphincterotome CleverCut2V)
  Other interventions: surgical intervention, endoscopic stenting, percutaneous transhepatic cholangiogram with balloon dilation
  Interventions: Procedure: Endoscopic sphincterotomy

INTERVENTIONS:
Procedure: Endoscopic papillary balloon dilation — treatment of endoscopic papillary balloon dilation
  Other Names: EPBD
  Arms: Endoscopic papillary balloon dilation
Procedure: Endoscopic sphincterotomy — treatment of endoscopic sphincterotomy
  Other Names: EST
  Arms: Endoscopic sphincterotomy

SUMMARY:
This study compares the effect of endoscopic sphincterotomy and endoscopic papillary balloon dilation in the treatment of acute biliary pancreatitis.Participants with acute biliary pancreatitis will be randomized into either the endoscopic sphincterotomy or endoscopic papillary balloon dilation groups.Moreover, the investigators compare the results obtained from the traditional bile/blood culture and metagenomics.

DETAILED DESCRIPTION:
Early endoscopic retrograde choledocho pancreatogram with endoscopic sphincterotomy is suggested in patients with acute biliary pancreatitis to reduce complication and mortality. Retrospective study of the investigators' hospital showed that endoscopic papillary balloon dilation is safe in the treatment of acute biliary pancreatitis. However, there is no report in literature concerning about the prospective study comparing the effect of endoscopic sphincterotomy and endoscopic papillary balloon dilation in the treatment of acute biliary pancreatitis.

Moreover, the presence of infective microorganisms in the biliary and/or pancreatic ducts may play important role in both the onset and outcome of acute biliary pancreatitis. Blood or bile obtained via endoscopic means is another way to know the causative bacterium/bacteria.

However, it still need considerable period of time to get the result of the culture. Recently, next-generation sequencing technologies have been developed, which can facilitate the analysis of a large number of microorganisms in different environments and human body sites. 16S(a svedberg unit) ribosomal deoxyribonucleic acid sequence analysis and metagenomics are two effective DNA sequencing approaches, and both have been used to study uncultivated gut microbial communities.

Aims:

1. To study the clinical effects of endoscopic sphincterotomy and endoscopic papillary balloon dilation in acute biliary pancreatitis.
2. To compare the results obtained from the traditional bile/blood culture and metagenomics.

Methods: Beginning from Jan 2016, patients with age ≥ 20 years and acute biliary pancreatitis concomitant with either signs of acute cholangitis or bile duct obstruction will be enrolled in the study. Participants will be randomized into either the endoscopic sphincterotomy or endoscopic papillary balloon dilation groups. The treatment effects and safety of both groups will be compared. The primary endpoint is the relative successful rates of retrieval of common bile duct stones of both groups. The secondary endpoint is the frequency of use of mechanical lithotripter, other drainage procedures, complication and mortality, as well as the number of treatment sections.

Besides blood culture exam, bile will be aspirated by placing a single-use, 5-French, standard catheter (after guide-wire cannulation) into the bile duct before the injection of contrast agent for endoscopic retrograde cholangiopancreaticography. Approximately 10 mL of bile will be collected and transferred in a sterile tube. Half of the bile obtained will be transported to the microbiology laboratory in blood culture bottles and in an anaerobic transport system. Bacteria will be cultured and identified according to the standard protocol used in our clinical microbiology laboratory. Another half of the bile specimen will be sending for metagenomic study. Finally, investigators will try to compare the results obtained from the traditional bile culture /blood culture and metagenomics, and to understand the effects of infective microorganisms in the biliary and/or pancreatic ducts on the acute biliary pancreatitis. In addition, investigators want to find out the best means of early and accurate diagnosis of the pathogen responsible for the infection.

ELIGIBILITY:
Patients with age ≥ 20 years and acute biliary pancreatitis concomitant with either signs of acute cholangitis or bile duct obstruction will be enrolled in the study. They will be randomized into two treatment groups (sphincterotomy vs. balloon dilation).

Inclusion Criteria:

Patients diagnosed with acute gallstone pancreatitis and fulfill any two items from a to c, plus one item in d, and e:

1. abdominal pain typical of pancreatitis;
2. elevation of serum amylase and/or lipase up to three times above normal;
3. imaging studies (abdominal ultrasound or abdominal computed tomography) showed evidence of pancreatitis
4. common bile duct stones, acute cholangitis (Charcot's triad), total bilirubin (total bilirubin)> 4mg / dL, bile duct dilatation (diameter> 6mm with intact gallbladder, or> 10mm when the gallbladder has been removed) plus total bilirubin 1.8 ~ 4mg / dL;
5. exclude other causes of acute pancreatitis.

Exclusion Criteria:

* septic shock
* serious coagulopathy (international normalized ratio 1.5, partial thromboplastin time greater than twice that of control, platelet count <50 x 1000 / Cumm)
* malignant tumors of the biliary and pancreatic tract
* severe cardiovascular or mental illness which can not cooperate with the exam and treatment;
* pregnant women
* patient who had ever received surgery or endoscopic treatment for biliopancreatic tract

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Complete removal of common bile duct stones | one year
  Successful bile duct clearance was defined as complete if the final cholangiogram revealed no more filling defects.

SECONDARY OUTCOMES:
Evaluation of adverse events | One week
  Adverse events were recorded according to the definitions and grading systems from the consensus of an American Society of Gastrointestinal Endoscopy Workshop. (P. B. Cotton, G. M. Eisen, L. Aabakken et al., "A lexicon for endoscopic adverse events: report of an ASGE workshop," Gastrointestinal Endoscopy, vol. 71, no. 3, pp. 446-454, 2010.)

CONTACTS AND LOCATIONS:
Overall Officials: Hoi Hung Chan, MD, PhD, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital., Kaohsiung City, Taiwan